CLINICAL TRIAL: NCT00970385
Title: Multicentric Study About Treatment of High Grade Peripheral T Cell Lymphoma in Adults. LTP Study Comparison Between VIP ABVD Versus CHOP
Brief Title: Study About Treatment of Newly Diagnosed Non Cutaneous Peripheral T Cell Lymphoma
Acronym: LTP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: French Innovative Leukemia Organisation (Other)
Responsible Party: CHU Grenoble/ Dr Rémy GRESSIN, GOELAMS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LTP 95
Record Dates: First submitted 2009-08-20; First posted 2009-09-02 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2009-09

CONDITIONS: Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — CHOP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CHOP 21 (Active Comparator): Induction therapy CHOP every 21 days:
  * cyclophosphamide 750 mg/m2 intravenously (IV) day 1
  * doxorubicin 50 mg/m2 IV day 1
  * vincristine 1,4 mg/m2 (maximum 2 mg) day 1
  * prednisone 100 mg/m2/D from D1 to D5.
  Interventions: Drug: CHOP21; Radiation: Radiotherapy consolidation
- VIP/ABVD arm (Experimental): VIP cycle:
  * etoposide 100 mg/m2/D IV from D1 to D3
  * ifosfamide 1000 mg/m2/D from D1 to D5
  * cisplatin 20 mg/m2/D as a continuous infusion from D1 to D5
  ABVD cycle:
  * doxorubicin50 mg/m2/D on D1 and D14
  * bleomycin 10 mg/m2/D
  * vinblastine 10 mg/m2/D
  * dacarbazine 375 mg/m2/D Each alternating cycle was repeated three times for a total of 6 cycles (3 VIP, 3 rABVD).
  Interventions: Drug: VIP/ABVD; Radiation: Radiotherapy consolidation

INTERVENTIONS:
Drug: CHOP21 — CHOP regimen:
  * cyclophosphamide 750 mg/m2 intravenously (IV) day 1
  * doxorubicin 50 mg/m2 IV day 1
  * vincristine 1,4 mg/m2 (maximum 2 mg) day 1
  * prednisone 100 mg/m2/D from D1 to D5.
  Other Names: CHOP 21 arm
  Arms: CHOP 21
Drug: VIP/ABVD — VIP regimen:
  * etoposide 100 mg/m2/D IV from D1 to D3
  * ifosfamide 1000 mg/m2/D from D1 to D5
  * cisplatinum 20 mg/m2/D as a continuous infusion from D1 to D5
  ABVD regimen:
  * doxorubicin50 mg/m2/D on D1 and D14
  * bleomycin 10 mg/m2/D
  * vinblastine 10 mg/m2/D
  * dacarbazine 375 mg/m2/D
  Other Names: VIP/ABVD Arm
  Arms: VIP/ABVD arm
Radiation: Radiotherapy consolidation — The treatment of Ann-Arbor stage I/II and stage III/IV patients with an initial bulky tumor (diameter ≥ 5 cm) was systematically completed by an irradiation plan. Forty grays were delivered (1,8 gray/day) over four weeks on the involved field.
  Other Names: Consolidation treatment

SUMMARY:
This is a multicenter randomized trial evaluating induction treatment with VIP-reinforced-ABVD (VIP-rABVD) versus CHOP/21 in patients with newly diagnosed peripheral T cell lymphoma.

DETAILED DESCRIPTION:
Induction therapy:

ARM 1: 6 Chemotherapy courses = 3 VIP alternated with 3 ABVD ARM 2: 8 Chemotherapy courses = CHOP every 21 days

Consolidation therapy:

For all patients if CR = radiotherapy 40GY / 5X1,8 GY per week

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed untreated PTCL
* age 18 and 70 years
* performance status ≤ 2
* Ann Arbor stage I to IV
* normal cardiac ventricular ejection fraction over 50%
* normal hepatic function (asat, ALAT, PAL < 2.5 ULN)

Exclusion Criteria:

* cutaneous form of PTCL
* previous treatment
* age < 18 and > 70
* performance status > 2
* abnormal cardiac or hepatic functions
* HIV-, HCV- or HBV- positivity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 1995-01; Primary Completion 2002-12 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Comparison between EFS rate of CHOP/21 versus VIP-rABVD in newly diagnosed PTCL. | 2 years

SECONDARY OUTCOMES:
Overall survival (OS) | 6 years
response rate at the end of the treatment | 6-8 months
progression free survival (PFS) | 6 years
hematotoxicity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Remy GRESSIN, MD MS, Principal Investigator — CHU Grenoble GOELAMS
Locations (1):
- Dr REMY GRESSIN, Grenoble, France